CLINICAL TRIAL: NCT00137657
Title: An Evaluation of the Impact of Cotrimoxazole Prophylaxis for HIV-Infected Adults on the Development of Antifolate Resistance Among Plasmodium Falciparum, Streptococcus Pneumoniae, and Escherichia Coli
Brief Title: Impact of Cotrimoxazole Prophylaxis for HIV-Infected Adults on Antifolate Resistance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: Kenya Medical Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: CDC-NCID-3354; UR6/CCU018970-02-2; SSC#664
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2005-12-13 (Estimated); Status verified 2005-08

CONDITIONS: HIV; Malaria; Diarrhea; Pneumonia; Opportunistic Infections
Keywords: HIV; malaria; E. Coli; S. pneumoniae; drug resistance; antifolate; opportunistic infections; Africa; Kenya; East Africa
MeSH Terms: conditions — Malaria; Diarrhea; Pneumonia; Opportunistic Infections; Escherichia coli Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

INTERVENTIONS:
Drug: Cotrimoxazole (trimethoprim sulfamethoxazole)

SUMMARY:
At least three studies in sub-Saharan Africa have demonstrated a decrease in morbidity or mortality among HIV-infected adults who took daily cotrimoxazole (trimethoprim sulfamethoxazole) [CTX] prophylaxis. Because of the demonstrated beneficial effect, high tolerability and low cost of CTX, the United Nations Programme on HIV/AIDS (UNAIDS) recommends that HIV-infected persons with symptomatic HIV or depressed CD4 counts receive daily CTX. The effect of this recommendation on subsequent development of antimicrobial resistance to antifolates among important pathogens needs to be evaluated. The investigators measured the change in the prevalence of markers of antifolate resistance among P. falciparum, and the change in the prevalence of CTX resistance among S. pneumoniae, and E. coli in HIV-infected individuals receiving CTX daily prophylaxis. In addition, the investigators measured the change in the prevalence of naso-pharyngeal or oro-pharyngeal carriage of CTX resistant S. pneumoniae among children living in households where an HIV-infected adult was receiving CTX daily prophylaxis.

DETAILED DESCRIPTION:
We conducted this study in Kisumu, Kenya where HIV prevalence is high and malaria is highly endemic. HIV infected and uninfected adults were assigned to receive daily CTX if CD4 cell count was <350, or daily multivitamin if CD4 cell count was >= 350 or if the client was HIV negative. All clients were then followed for a total of 6 months. At specified scheduled and sick visits, clients received a physical exam, blood smears, nasopharyngeal swabs and stool samples or rectal swabs. Samples collected at baseline and during follow-up were used to measure the change in CTX resistance among P. falciparum parasites, pneumococcus isolates, and commensal E. coli.

ELIGIBILITY:
Inclusion Criteria:

Clients presenting to the CRC HIV counseling and testing site in Kisumu were eligible for the study if they met the following inclusion criteria:

* 15 years of age or older
* Able to make all follow-up visits (i.e. do not plan to leave Kisumu during the next 6 months, are not homebound)
* Able to understand and give informed consent.

Exclusion Criteria:

Clients were not eligible for the study if they met any of the following exclusion criteria:

* Known allergic reaction to sulfa medications (i.e. CTX, sulfadoxine- pyrimethamine)
* Women in their first trimester of pregnancy or planning to become pregnant in the next 6 months
* Clients taking daily antibiotics for treatment of a chronic illness; or prophylaxis, excluding tuberculosis treatment.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1478
Dates: Start 2002-02; Study Completion 2003-11

PRIMARY OUTCOMES:
Change in Plasmodium falciparum molecular markers of antifolate resistance before and while taking daily CTX
Change in nasopharyngeal pneumococcal resistance before and while taking daily CTX, and among children living in households where adults are taking daily CTX
Change in commensal E. coli resistance before and while taking daily CTX

SECONDARY OUTCOMES:
To measure CTX-resistance among Salmonella and other enteric bacterial pathogens in patients with diarrhea in the study area
To assess the efficacy of sulfadoxine-pyrimethamine (SP) treatment of breakthrough P. falciparum parasitemia and clinical malaria among HIV-infected persons taking daily CTX prophylaxis
To measure sulfa metabolite levels in HIV-infected persons receiving daily CTX who develop a drug reaction, to determine if differing rates of metabolism contribute to the development of adverse reactions
To assess the effect of daily CTX prophylaxis on the etiology of diarrheal diseases in HIV-infected persons
To evaluate the serotype distribution of and immune response to colonizing pneumococci
To assess the cause of diarrheal diseases among HIV-infected persons
To measure the change in quality of life indicators among clients receiving daily CTX

CONTACTS AND LOCATIONS:
Overall Officials: Mary J Hamel, M.D., Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- CDC KEMRI Research Institute, Kisumu, Kenya